CLINICAL TRIAL: NCT06955806
Title: Clinical Efficacy and Molecular Dynamics of Quantum Molecular Resonance (QMR) Electrotherapy in Dry Eye Management
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSE Sung Hei Jimmy, Assistant Professor of Practice, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HSEARS20250209003
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye Disease (DED)
Keywords: Dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Active Comparator): Following a comprehensive evaluation, the treatment group will undergo a 20-minute treatment once per week for four weeks.
  Interventions: Device: The Rexon-Eye, an electrotherapy device utilizing Quantum Molecular Resonance (QMR) technology
- Control Arm (Sham Comparator): Following a comprehensive evaluation, the sham treatment group will firstly undergo a 20-minute sham treatment once per week for four weeks. Two additional comprehensive evaluations and tear fluid collections will be conducted one month and three months after the completion of the treatment period.
  After the three-month post-treatment evaluation, the control group will receive four weekly treatments.
  Interventions: Device: The Rexon-Eye, an electrotherapy device utilizing Quantum Molecular Resonance (QMR) technology

INTERVENTIONS:
Device: The Rexon-Eye, an electrotherapy device utilizing Quantum Molecular Resonance (QMR) technology — The device has received EC certification as a medical device for the treatment of ocular surface disorders. It will deliver a low-intensity alternating electrical current (ranging from 4 MHz to 64 MHz) to targeted biological tissue via contact electrodes. Previous studies have shown the effectiveness of this treatment in alleviating dry eye symptoms, both subjectively and objectively.

SUMMARY:
This project aims to investigate the clinical efficacy and molecular mechanisms of Quantum Molecular Resonance (QMR) electrotherapy in the management of dry eye disease (DED). DED is a multifactorial condition characterized by tear film instability, hyperosmolarity, inflammation, and neurosensory abnormalities, leading to discomfort and visual disturbances. The Rexon-Eye device, which utilizes QMR technology, has shown positive effects in alleviating dry eye symptoms. However, the exact mechanisms by which the stimulation of high-frequency electrical fields promotes improvement in DED remain unclear.

The research will be conducted as a longitudinal study involving 30 participants between the ages of 18 and 40 who meet the diagnostic criteria for DED. Participants will be randomly assigned to either a treatment group receiving QMR electrotherapy or a control group receiving a sham treatment, followed by a real treatment after second evaluation. Each participant in the treatment group will undergo a 20-minute weekly session for four weeks, with clinical evaluations and tear fluid collection occurring throughout the study.

Comprehensive assessments will be performed to evaluate tear film stability, lipid layer composition, ocular surface health and corneal sensitivity. Tear samples collected during the study will undergo molecular analysis using mass spectrometry to identify biochemical changes associated with QMR electrotherapy. Additionally, safety evaluations will be conducted at each visit to monitor potential adverse effects.

The study aims to determine whether QMR electrotherapy effectively improves clinical dry eye parameters while also uncovering the molecular changes in tear composition that may underlie its therapeutic effects. By exploring both clinical outcomes and biological mechanisms, this research will contribute valuable insights into the potential of QMR electrotherapy as an innovative treatment for dry eye disease.

DETAILED DESCRIPTION:
Study Purpose and Potential Benefits:

Recently, a high frequency electrotherapy device using Quantum Molecular Resonance (QMR) technique, the Rexon-Eye was being developed for dry eye treatment. During the treatment, a low-intensity, high-frequency (a spectrum of frequencies ranging from 4 MHz to 64 MHz) electrical stimulations are applied on the epidermis of closed eyelids up to the lid border by specially designed goggles. Previous data showed that it could effectively improve symptoms and clinical signs of DED by increasing the tear secretion and improving the meibomian gland function. Compared with conventional DED management options such as lubricant and warm compress, previous studies proposed that this treatment may allow a possible capability to induce reactivation of physiological lacrimal functions instead of a short-term symptom relief.

The aims of this project are to investigate the clinical efficacy of QMR electrotherapy and the associated changes in tear proteomics and lipidomics in the management of dry eye disease.

Participant Eligibility

* aged 18 to 40 years old
* with habitual or best corrected visual acuity better than or equal to 6/9
* diagnosed as dry eye disease according to OSDI score (13 or above) and at least one positive result from dry eye assessment.

Exclusion criteria:

* history of ocular inflammation, trauma or surgery within 6 months
* long-term ocular medications
* current dry eye treatment
* uncontrolled, newly diagnosed systemic diseases
* with modified long-term medications within 6 months that are known to affect tear profile
* carrying active implantable devices (e.g., pacemakers and hearing aids) Contact lens wearers will be required to stop contact lens wear 1 month before the first evaluation and during the whole study period.

Study Procedure All the participants will be given a comprehensive dry eye assessment at the baseline visit (visit1). The assessment includes questionnaire filling, ocular surface checking, tear fluid examination and collection, and eyelid examination.

Participants will then be assigned to receive QMR treatment, which requires four sessions of treatment (on a weekly basis). Two post treatment comprehensive dry eye assessment will be scheduled one month after the 4th treatment, and three months after the 4th treatment.

Some participants may be given another four sessions of treatment (on a weekly basis), followed by two post treatment comprehensive dry eye assessment (also one month after the 4th treatment, and three months after the 4th treatment). In summary, some participants need to visit us 6 times in 5 months while the others may need to visit us 12 times in 8 months.

Parameters to be assessed in Comprehensive evaluation:

* Dry Eye Disease (DED) questionnaires - Ocular Surface Disease Index (OSDI)
* Non-invasive tear break-up time (NITBUT), tear meniscus height (TMH) - Keratograph® 5M
* Lipid layer thickness (LLT) and infrared meibography - idra® Ocular Surface Analyser
* External ocular health, ocular surface staining and lid margin assessment - Slit-lamp biomicroscopy and fluorescein strips
* Corneal sensitivity - Corneal Esthesiometer Brill

Potential Risk(s) or Discomfort(s) and their minimization(s):

EC certificate has certified the device safety of Rexon-Eye including electrical safety and electromagnetic compatibility, and also its clinical safety and effectiveness in treating DED. There is no anticipated risk to participants according to the current literature. All procedures will be conducted by a registered or student optometrist.

Some possible treatment induced effects included a sensation of about 3 to 4°C temperature increment underneath the treatment goggles; transient blurred vision after treatment caused by the pressure of the goggles to the closed eyelid; or transient eyelid skin redness for subjects with sensitive skin. From published results, all these effects should be reversible and disappear within minutes after the treatment is finished. Eye check will be done before and after the treatment to avoid any potential problem.

The treatment will be terminated if the subject is sensitive to the procedure or any unexpected adverse response is observed during the study.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 40 years old
* with habitual or best corrected visual acuity better than or equal to 6/9
* diagnosed as dry eye disease according to OSDI score (13 or above) and at least one positive result from dry eye assessment.

Exclusion Criteria:

* history of ocular inflammation, trauma or surgery within 6 months
* long-term ocular medications
* current dry eye treatment
* uncontrolled, newly diagnosed systemic diseases
* with modified long-term medications within 6 months that are known to affect tear profile
* carrying active implantable devices (e.g., pacemakers and hearing aids)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical efficacy | From enrollment to the end of treatment at 4 (Treatment group) to 8 (Sham treatment group)months
  Ocular Surface Disease Index

SECONDARY OUTCOMES:
The associated tear proteomics and lipidomics changes after Electrotherapy | From enrollment to the end of treatment at 4 (Treatment group) to 8 (Sham treatment group)months
  The associated changes in tear proteomics and lipidomics will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trivli A, Karmiris E, Dalianis G, Ruggeri A, Terzidou C. Evaluating the efficacy of Quantum Molecular Resonance (QMR) electrotherapy in mixed-type dry eye patients. J Optom. 2023 Apr-Jun;16(2):128-134. doi: 10.1016/j.optom.2022.06.003. Epub 2022 Jul 16. PMID 35851496